CLINICAL TRIAL: NCT01864889
Title: Clinical Study of Chimeric CD(Cluster of Differentiation)19 Antigen Receptor-modified T Cells in Relapsed and/or Chemotherapy Refractory B-cell Leukemias and Lymphomas
Brief Title: Treatment of Relapsed and/or Chemotherapy Refractory B-cell Malignancy by CART19
Acronym: CART19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-005
Record Dates: First submitted 2013-05-20; First posted 2013-05-30 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CD19 CAR T cells (Experimental): Patients receive anti-CD19-CAR retroviral vector-transduced autologous or donor-derived T cells on days 0,1, 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-CD19-CAR vector-transduced T cells

INTERVENTIONS:
Biological: anti-CD19-CAR vector-transduced T cells — genetically engineered lymphocyte therapy
  Other Names: genetically engineered lymphocyte therapy

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is studying genetically engineered lymphocyte therapy in treating patients with B-cell leukemia or lymphoma that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD19 (cluster of differentiation antigen 19 ) vector (referred to as CART-19 cells).

II. Determine duration of in vivo survival of CART-19 cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of CART-19 TCR (T-cell receptor) zeta:CD137 and TCR zeta cells over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-tumor response due to CART-19 cell infusions.

II. To determine if the CD137 transgene is superior to the TCR zeta only transgene as measured by the relative engraftment levels of CART-19 TCR zeta:CD137 and TCR zeta cells over time.

III. Estimate relative trafficking of CART-19 cells to tumor in bone marrow and lymph nodes.

IV. For patients with stored or accessible tumor cells (such as patients with active chronic lymphocytic leukemia(CLL), acute lymphocytic leukemia (ALL), etc) determine tumor cell killing by CART-19 cells in vitro.

V. Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable CART-19 (loss of engraftment).

VI. Determine the relative subsets of CART-19 T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment.

Patients receive anti-CD19-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on days 0,1, and 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled

  * CD19+ leukemia or lymphoma
  * ALL in CR2(second complete remission) or CR3(third complete remission) and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor
  * Follicular lymphoma, previously identified as CD19+:
  * At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy
  * Stage III-IV disease
  * Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year)
  * Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)
  * CLL:
  * At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy. Patients with high risk disease manifested by deletion chromosome 17p will be eligible if they fail to achieve a CR to initial therapy or progress within 2 years of 1 prior
  * Less than 2 years between last chemotherapy and progression (i.e. most recent progression free interval < 2 years)
  * Not eligible or appropriate for conventional allogeneic SCT
  * Patients who achieve only a partial response to FCR(fludarabine, cyclophosphamide and Rituxan) as initial therapy will be eligible.
  * Mantle cell lymphoma:
  * Beyond 1st CR (complete remission) with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
  * Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc...)
  * Relapsed after prior autologous SCT
  * B-cell prolymphocytic leukemia (PLL) with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT
  * Diffuse large cell lymphoma, previously identified as CD19+:
  * Residual disease after primary therapy and not eligible for autologous SCT
  * Relapsed after prior autologous SCT
  * Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate of conventional allogeneic or autologous SCT
  * Expected survival > 12 weeks
  * Creatinine < 2.5 mg/dl
  * ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal
  * Bilirubin < 2.0 mg/dl
  * Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy
  * Adequate venous access for apheresis, and no other contraindications for leukapheresis
  * Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women

  * The safety of this therapy on unborn children is not known
  * Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
  * Uncontrolled active infection
  * Active hepatitis B or hepatitis C infection
  * Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
  * Previously treatment with any gene therapy products
  * Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation
  * Any uncontrolled active medical disorder that would preclude participation as outlined
  * HIV infection

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-tumor responses to CART-19 cell infusions | up to 24 weeks

OTHER OUTCOMES:
in vivo existence of CART19 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang WY, Liu Y, Wang Y, Nie J, Guo YL, Wang CM, Dai HR, Yang QM, Wu ZQ, Han WD. Excessive activated T-cell proliferation after anti-CD19 CAR T-cell therapy. Gene Ther. 2018 Jun;25(3):198-204. doi: 10.1038/s41434-017-0001-8. Epub 2018 Mar 29. PMID 29599530
- [Derived] Dai H, Zhang W, Li X, Han Q, Guo Y, Zhang Y, Wang Y, Wang C, Shi F, Zhang Y, Chen M, Feng K, Wang Q, Zhu H, Fu X, Li S, Han W. Tolerance and efficacy of autologous or donor-derived T cells expressing CD19 chimeric antigen receptors in adult B-ALL with extramedullary leukemia. Oncoimmunology. 2015 May 26;4(11):e1027469. doi: 10.1080/2162402X.2015.1027469. eCollection 2015 Nov. PMID 26451310